CLINICAL TRIAL: NCT07267728
Title: A Clinical Study to Assess the Effect of a Dietary Supplement on Menstrual Cycle Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muse Nutrition Ltd (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20736
Record Dates: First submitted 2025-11-19; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Premenstrual Syndrome; Menstrual Pain
Keywords: Bloating; Mood Disorders
MeSH Terms: conditions — Premenstrual Syndrome; Dysmenorrhea; Mood Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DITTO Cycle Supplement (Experimental): Participants will take two capsules of the DITTO Cycle Supplement once daily, starting two days after menstrual bleeding ends, for the duration of three menstrual cycles.
  Interventions: Dietary Supplement: DITTO Cycle Supplement

INTERVENTIONS:
Dietary Supplement: DITTO Cycle Supplement — The capsules should be taken in the morning with the first meal and a glass of water.

SUMMARY:
This is a single-group, virtual clinical trial evaluating the effects of a daily dietary supplement (DITTO Cycle Supplement) on menstrual cycle symptoms across three menstrual cycles. The study investigates changes in symptom severity and quality of life through validated questionnaires including the Menstrual Symptoms Questionnaire (MSQ).

ELIGIBILITY:
Inclusion Criteria:

* Female-at-birth
* Aged 18-45
* In the last three menstrual cycles, has experienced three or more of the following symptoms associated with their menstrual cycle: Menstrual cramps, Bloating, Breast tenderness, Headaches, Fatigue, Muscle aches and/or joint pain, Cravings, Mood swings, Low mood, Feelings of anxiety, Irritability, Difficulty concentrating
* Generally healthy - does not live with any uncontrolled chronic disease
* Has a regular menstrual cycle length, between 23 and 35 days
* Tracks their menstrual cycle and can predict their period dates
* Anyone willing to comply with study requirements
* Anyone with no known allergies to the ingredients listed in the product

Exclusion Criteria:

* Anyone with pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders
* Women who are pregnant, breastfeeding, or trying to conceive
* Anyone unwilling to follow the study protocol
* Anyone in perimenopause, menopause, or experiencing menopausal-type symptoms
* Anyone with planned surgery during the study period
* Anyone with a history of substance abuse
* Anyone diagnosed with high blood pressure, high cholesterol, heart disease, heart attack, stroke, irregular heartbeat (AFib), clogged arteries, poor circulation, heart failure, or other heart conditions
* Anyone diagnosed with a hormone or reproductive health-related cancer or benign condition
* Anyone diagnosed with a menstrual health condition such as endometriosis, PCOS, or adenomyosis
* Anyone diagnosed with diabetes or other endocrine-related condition
* Anyone currently participating or planning to participate in a research study
* Anyone who has started, changed, or stopped taking hormonal birth control in the last three months
* Has a planned insertion or replacement of an IUD in the next 12 weeks

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Menstrual Symptoms Questionnaire (MSQ) Scores | Baseline, End of Cycle 1(28 days), End of Cycle 2(28 days), End of Cycle 3 (28 days)
  Change from baseline in menstrual symptom severity as measured by the Menstrual Symptoms Questionnaire (MSQ), including cramps, bloating, fatigue, mood swings, breast tenderness, headaches, anxiety, irritability, and difficulty concentrating.

SECONDARY OUTCOMES:
Change in Menstrual-Related Quality of Life | Baseline, End of Cycle 1(28 days), End of Cycle 2(28 days), End of Cycle 3 (28 days)
  Change from baseline in participant-reported quality of life related to menstrual symptoms, measured using study-specific self-report questionnaires evaluating overall impact on daily living and well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Las Vegas, Nevada, United States